CLINICAL TRIAL: NCT07056751
Title: The Effects of Artificial Air Negative Ions on High-Altitude Acclimatization
Brief Title: The Effects of Artificial Air Negative Ions on High-Altitude Acclimatization, Serum HIF1, and PWC170 Index
Acronym: 2022JW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Putian City, Putian, Fujian (Other Government)
Responsible Party: Principal Investigator, Zhizhong Chen, Doctor, The First Hospital of Putian City, Putian, Fujian
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FirstHPCF
Record Dates: First submitted 2025-06-22; First posted 2025-07-09 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Negative Air Ions; Altitude Sickness; High-altitude Adaptation
Keywords: Air negative ions; High-Altitude Adaptation; high-altitude reactions; PWC170
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Air negative ion intervention study (Experimental): Arm 1: observation group (air negative ion intervention group) consisting of 30 individuals
  Interventions: Device: Air negative ion intervention study
- No air negative ion intervention (Placebo Comparator): Arm 2: control group (no air negative ion intervention group) consisting of 30 individuals
  Interventions: Device: No air negative ion intervention

INTERVENTIONS:
Device: Air negative ion intervention study — The observation group received air negative ion intervention every night for one week before entering the plateau (from 22:00 to 06:00). Before entering the plateau, they were in Putian City, China, where the temperature was about 28°C, humidity was about 68%, and the concentration of negative ions was approximately 800/cm³. The air negative ion converter used was the Mi Energy ET-21 model from RELTEC Medical Devices Corporation. Air negative and positive ion concentrations were measured using an ion detector (NKMH-103, HOKUTO, Japan) to ensure that each participant's room had a negative ion concentration of around 100,000/cm³.
  Arms: Air negative ion intervention study
Device: No air negative ion intervention — No air negative ion intervention
  Arms: No air negative ion intervention

SUMMARY:
To explore the effects of negative ions generated by an ion converter on the high-altitude acclimatization of healthy populations and their impact on serum HIF1 (hypoxia-inducible factor 1) and PWC170 index after entering high-altitude areas.

DETAILED DESCRIPTION:
Objective: To explore the effects of negative ions generated by an ion converter on the high-altitude acclimatization of healthy populations and their impact on serum HIF1 and PWC170 index after entering high-altitude areas.

Methods: Sixty healthy adults were randomly divided into two groups: an air negative ion intervention group (observation group) of 30 participants and a non-air negative ion intervention group (control group) of 30 participants. Air negative ion intervention was conducted one week before entering high-altitude areas, lasting for 8 hours each day. Before entering high-altitude areas, measurements were taken for height, weight, blood pressure, heart rate, routine blood tests, routine urine tests, biochemical profiles, blood oxygen saturation, and HIF1 (hypoxia-inducible factor 1). One week after entering high-altitude areas, the above indicators were retested, and the PWC170 index was calculated to evaluate changes in endurance during high-altitude activities.

ELIGIBILITY:
Inclusion Criteria:

healthy non-smoking men aged 18 or above and long-term residents of the plains no history of high-altitude exposure in the past 6 months no cardiovascular or pulmonary diseases not currently taking any medications.

Exclusion Criteria:

Tibetan ethnicity long-term residents of high altitudes history of high-altitude exposure in the past 6 months currently taking cold medicine, vitamins, corticosteroids, or other drugs presence of acute or chronic illnesses

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
High-Altitude Acclimatization | two weeks
  Following their ascent to high altitudes, all participants completed the Acute Mountain Sickness (AMS) questionnaire daily, with AMS diagnosis based on the Lake Louise Criteria.

SECONDARY OUTCOMES:
PWC170 Index | one day
  This study employed a two-stage quantitative load stepping exercise. The first stage involved stepping at a height of 30cm, a speed of 24 steps/min, and a duration of 4 minutes. After a 4-minute rest, the second stage was performed with the same step height and duration as the first stage but at a speed of 35 steps/min controlled by a metronome. Power and PWC170 were calculated using the following formulas: Power (Kg · m / min) = 4/3 [Body weight (Kg) × Step height (m) × Total number of step-ups and step-downs (b/min)] PWC170 (Kg · m / min) = N1 + (N2 - N1) [(170 - f1) / (f2 - f1)] Where N1 and N2 represent the power in the first and second stage loads, and f1 and f2 are the immediate pulse rate at the first and second stage loads (b/min).

CONTACTS AND LOCATIONS:
Locations (1):
- The Ethics Committee of Putian 95 Hospital, Putian, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 07.01.2025-no end date
Access Criteria: Scientific researcher
URL: https://register.clinicaltrials.gov/prs/beta/studies/S000FYQ700000078/protocol/ipdSharing?edit=true